CLINICAL TRIAL: NCT07405892
Title: The Impact of Hypotension Prediction Index-Guided Management on Intraoperative Hypotension and Major Postoperative Complications in Patients Undergoing Oral Cancer Resection and Reconstruction
Brief Title: Applying HPI in Oral Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202507237RINB
Record Dates: First submitted 2026-01-21; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: the Severity and Duration of Intraoperative Hypotension
Keywords: intraoperative hypotension

STUDY DESIGN:
Intervention Model Description: intervention: HPI guidance; control: HPI silence
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were blinded to their group allocation, and outcome assessors were also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI (Experimental): HPI guidance
  Interventions: Device: HPI
- HPI silence (Active Comparator): HPI silence
  Interventions: Device: HPI silence

INTERVENTIONS:
Device: HPI — HPI guidance for intraoperative hypotension management
  Arms: HPI
Device: HPI silence — No HPI guidance for intraoperative hypotension management
  Arms: HPI silence

SUMMARY:
Investigating HPI effect in oral cancer surgery

DETAILED DESCRIPTION:
Intraoperative hypotension, defined as a mean arterial pressure (MAP) below 65 mmHg, is common during oral cancer resection with reconstruction-a lengthy procedure averaging 13 hours. Prolonged anesthesia increases the risk of intraoperative hypotension, which would lead to a higher need for vasopressor administration and fluid transfusion. Additionally, surgical anastomosis sites are vulnerable, and hypotension has been linked to increased risks of anastomotic necrosis, septic shock, organ failure, and mortality.

The Hypotension Prediction Index (HPI) is a machine-learning-based algorithm introduced in 2019 that analyzes arterial pressure waveform characteristics to provide real-time monitoring and early prediction of hypotensive episodes-defined as a MAP <65 mmHg lasting for at least one minute-during surgery. Recent randomized controlled trials have evaluated the effectiveness of HPI-guided management in preventing intraoperative hypotension. These studies commonly use the "time-weighted average (TWA) MAP <65 mmHg" as the primary outcome, calculated as the area under the threshold (in mmHg×hours) divided by the total duration of surgery (in hours). The lower the value, the shorter and less severe the intraoperative hypotension. However, limited studies have specifically investigated the impact of HPI-guided management on the duration and severity of intraoperative hypotension and postoperative complications in patients undergoing oral cancer resection with reconstruction.This study aims to evaluate the effectiveness of HPI-guided management in reducing the duration and severity of intraoperative hypotension in patients undergoing oral cancer resection with free flap reconstruction. The investigator hypothesize that the TWA-MAP <65 mmHg will be significantly lower in the HPI-guided group compared to the standard care group. Postoperative major complications will be followed during postoperative 30 days. One hundred patients aged 20 to 80 years undergoing elective oral cancer resection with free flap reconstruction will be randomized to receive hemodynamic management with or without HPI guidance. Clinicians caring for patients assigned to the HPI guidance group will be alerted when the index exceeded 85 (range 0 to 100) indicating the later occurrence of MAP< 65mmHg for at least minutes and a treatment protocol based on advanced hemodynamic parameters recommended vasopressor or inotrope, fluid administration, or observation. Primary outcome is the data of TWA-MAP<65mmHg. Postoperative complications and mortality will be followed up to postoperative 30 days.

ELIGIBILITY:
Inclusion Criteria:

* elective oral cancer surgery with free flap reconstruction

Exclusion Criteria:

* severe arrhythmia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
time weight average mean arterial pressure less than 65 mmHg | the duration of surgery
  a value indicating the severity and duration of intraoperative hypotension

IPD SHARING:
Plan to Share IPD: No
due to ethical concern